CLINICAL TRIAL: NCT04767191
Title: Efficacy of Artemether Lumefantrine (AL) and Dihydroartemisinin-Piperaquine (DHP) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Siaya and Bungoma Counties, Kenya
Brief Title: Malaria Therapeutic Efficacy Study (TES) Kenya
Acronym: Kenya-TES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Kenya Ministry of Health (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012257
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Uncomplicated Malaria
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: The two drugs being assessed are already approved and in use by the Kenya Ministry of Health as the 1st and 2nd line treatments for malaria. The study is to assess the continued efficacy of the drugs.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artemether lumefantrine (Active Comparator): The drug is approved and in use by the Kenya Ministry of Health as the 1st line treatment for malaria. The study is to assess the continued efficacy of the drug.
  Interventions: Drug: artemether lumefantrine
- dihydroartemisinin piperaquine (Active Comparator): The drug is approved and in use by the Kenya Ministry of Health as the 2nd line treatment for malaria. The study is to assess the continued efficacy of the drug.
  Interventions: Drug: dihydroartemisinin piperaquine

INTERVENTIONS:
Drug: artemether lumefantrine — The drugs are approved and in use by the Kenya Ministry of Health as the 1st and 2nd line treatment for malaria. The study is to assess the continued efficacy of the two drugs in the treatment of uncomplicated malaria.
  Arms: artemether lumefantrine
Drug: dihydroartemisinin piperaquine — Antimalarial Combinations
  Arms: dihydroartemisinin piperaquine

SUMMARY:
WHO recommends that Therapeutic Efficacy Studies (TES) for 1st and 2nd line antimalarial medicines should be routinely carried out and data made available for decision-making due to the threat of emergence and spread of artemisinin resistance in malaria-endemic countries, especially in Africa. In line with this WHO recommendation, Kenya Ministry of Health (MOH) is conducting the TES to determine the efficacy of artemether lumefantrine (AL), and dihydroartemisinin-piperaquine (DHP), the first and second line treatment of uncomplicated malaria in Kenya. The objective of this study is to inform the decisions or actions made by a public health authority (Kenya Ministry of Health) to inform decision on revision of the antimalarial guidelines and policy in Kenya. Jhpiego's Impact Malaria project in Kenya, with funding and technical oversight from US President's Malaria Initiative (PMI) through USAID and CDC, will support the Kenya MOH in its effort to evaluate the efficacy of AL and DHP in the treatment of children with uncomplicated malaria. The study is being conducted by Kenya MOH, with technical support and funding by PMI-USAID through Jhpiego in Kenya.

DETAILED DESCRIPTION:
WHO recommends that Therapeutic Efficacy Studies (TES) for 1st and 2nd line antimalarial medicines should be routinely carried out and data made available for decision-making due to the threat of emergence and spread of artemisinin resistance in malaria-endemic countries, especially in Africa. In its strategy to strengthen malaria surveillance, Kenya's Ministry of Health (MOH) National Malaria Program (NMP) planned to conduct TES every three years to ascertain continuing efficacy of the first and second-line treatments. The last TES for 1st line treatment of malaria in Kenya was done in Siaya county in 2016. In line with the WHO recommendation, Jhpiego Impact Malaria project in Kenya, with funding and technical oversight from Center for Disease Prevention and Control (CDC) will be supporting the Kenya MOH NMP to conduct a TES to assess the efficacy of the current first and second line treatment policy in Kenya. The study is being conducted by Kenya MOH NMP, with technical oversight and funding by CDC through the Jhpiego Impact Malaria project in Kenya.

Objective: To assess the efficacy of Artemether Lumefantrine (AL) and Dihydroartemisinin-Piperaquine (DHP) for the treatment of uncomplicated P. falciparum malaria infections.

Study Sites: One site will be selected in Siaya county and one site will be selected in Bungoma county (Kimilili Sub-County). Both sites will be Level-2 facilities (health centers) with high outpatient department attendance of patients with malaria. At each site, there will be two study arms: one arm for AL and one arm for DHP.

Study Period: March 2021 to September 2021

Study Design: This surveillance study is a two-arm prospective study Patient population: Febrile patients aged between 6 months and 59 months, with confirmed uncomplicated P. falciparum monoinfection.

Sample Size: At each site, at least 100 patients will be enrolled per drug (200 patients per site, 400 patients total).

Treatment(s) and follow-up: Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate AL efficacy, and over a 42-day follow-up period to evaluate DHP efficacy.

Primary endpoints: The proportion of patients with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response as indicators of efficacy. Recrudescence will be distinguished from re-infection by polymerase chain reaction (PCR) analysis.

Secondary endpoints: The frequency and nature of adverse events.

Exploratory endpoints: to determine the polymorphism of molecular markers of drug resistance and evasion of diagnostic testing; to determine the blood concentration of AL

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months to 59 months; mono-infection with P. falciparum confirmed by positive blood smear (i.e. no mixed infection);
* parasitaemia of 1,000 - 100,000/µl asexual forms;
* presence of axillary temperature ≥ 37.5 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* haemoglobin ≥5.0 g/dL at admission;
* informed consent from a parent or guardian;
* parent/guardian agrees to bring the patient for planned follow-up visits at day 7, 14, 21, and 28

Exclusion Criteria:

* general danger signs or signs of severe falciparum malaria according to the definitions of WHO;
* severe malnutrition according to WHO child growth standards (WHO, 2006), children with marasmus or oedematous malnutrition;
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s);
* history of receiving any antimalarial treatment in the preceding 72 hours;. exposure to malaria vaccine

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Number of patients (in the Artemether Lumefantrine arm) with clinical and parasitological cure (i.e. free of malaria symptoms and parasites) assessed clinically and via microscopy and rapid diagnostic test. | By day 28 post-treatment
Number of patients (in the Dihydroartemisinin-Piperaquine arm) with clinical and parasitological cure (i.e. free of malaria symptoms and parasites) assessed clinically and via microscopy and rapid diagnostic test. | By day 42 post-treatment

SECONDARY OUTCOMES:
Number of patients (in the Artemether Lumefantrine arm arm) with treatment-related adverse events | by day 28 post-treatment
Number of patients (in the Dihydroartemisinin-Piperaquine arm) with treatment-related adverse events | by day 42 post-treatment
Number of patients (in the Artemether Lumefantrine arm) with molecular markers of drug resistance assessed via phenotype test | by day 28 post-treatment
Number of patients (in the Dihydroartemisinin-Piperaquine arm) with molecular markers of drug resistance assessed via phenotype test | by day 42 post-treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Makhonge Health Centre, Bungoma, Bungoma County
  - Kaluo Health Centre, Siaya, Siaya County

IPD SHARING:
Plan to Share IPD: No